CLINICAL TRIAL: NCT05693649
Title: Behavioral Economic Approaches for Population-Based Colorectal Cancer Screening
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Principal Investigator, Shivan Mehta, Principal Investigator, Abramson Cancer Center at Penn Medicine
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Screening
Other Study IDs: UPCC 14022
Record Dates: First submitted 2023-01-12; First posted 2023-01-23 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Cancer
Keywords: Prevention; Cancer Screening; Behavioral Economics
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Arm 1A: Usual Care (Experimental): Patients assigned to the Usual Care arm will receive current usual care and will not receive direct patient outreach or any visit-based interventions from this trial.
  Interventions: Behavioral: No Direct Patient Outreach; Behavioral: No Nudge/Text
- Arm 2A: Colonoscopy Only and No Nudge/Text (Experimental): Using bulk ordering, patients assigned to this arm will receive an order for colonoscopy and direct outreach (via text message and either the electronic patient portal or mailed letter, depending on their patient portal status) informing them they are overdue for CRC screening. Patients randomized to this arm will not receive visit-based interventions.
  Interventions: Behavioral: Direct Patient Outreach: Colonoscopy Only; Behavioral: No Nudge/Text
- Arm 2B: Colonoscopy Only and Visit-Based Nudge/Text (Experimental): Using bulk ordering, patients assigned to this arm will receive an order for colonoscopy and direct outreach (via text message and either the electronic patient portal or mailed letter, depending on their patient portal status) informing them they are overdue for CRC screening. Patients randomized to this arm who attend a visit with their Primary Care Physician (PCP) will additionally receive a visit-based, clinician directed nudge to discuss colorectal cancer screening and a follow-up text 3 days post-visit to encourage screening completion.
  Interventions: Behavioral: Direct Patient Outreach: Colonoscopy Only; Behavioral: Visit-Based Nudge/Text
- Arm 3A: Sequential Choice and No Nudge/Text (Experimental): Using bulk ordering, patients assigned to this arm will receive an order for colonoscopy and direct outreach (via text message and either the electronic patient portal or mailed letter, depending on their patient portal status) informing them they are overdue for CRC screening. If not completed, patients will receive an order and a mailed fecal immunochemical test (FIT) with a reminder to complete CRC screening. Patients randomized to this arm will not receive visit-based interventions.
  Interventions: Behavioral: Direct Patient Outreach: Sequential Choice; Behavioral: No Nudge/Text
- Arm 3B: Sequential Choice and Visit-Based Nudge/Text (Experimental): Using bulk ordering, patients assigned to this arm will receive an order for colonoscopy and direct outreach (via text message and either the electronic patient portal or mailed letter, depending on their patient portal status) informing them they are overdue for CRC screening. If not completed, patients will receive an order and a mailed fecal immunochemical test (FIT) with a reminder to complete CRC screening. Patients randomized to this arm who attend a visit with their Primary Care Physician (PCP) will additionally receive a visit-based, clinician directed nudge to discuss colorectal cancer screening and a follow-up text 3 days post-visit to encourage screening completion.
  Interventions: Behavioral: Direct Patient Outreach: Sequential Choice; Behavioral: Visit-Based Nudge/Text

INTERVENTIONS:
Behavioral: No Direct Patient Outreach — Patient will not receive direct outreach prompting them to schedule and/or complete colorectal cancer screening.
  Arms: Arm 1A: Usual Care
Behavioral: Direct Patient Outreach: Colonoscopy Only — Patient will receive direct outreach including an order to schedule and complete colonoscopy.
  Arms: Arm 2A: Colonoscopy Only and No Nudge/Text; Arm 2B: Colonoscopy Only and Visit-Based Nudge/Text
Behavioral: Direct Patient Outreach: Sequential Choice — Patient will receive direct outreach including an order to schedule and complete colonoscopy then an at-home fecal immunochemical test (FIT) if colonoscopy is not completed.
  Arms: Arm 3A: Sequential Choice and No Nudge/Text; Arm 3B: Sequential Choice and Visit-Based Nudge/Text
Behavioral: Visit-Based Nudge/Text — Patient's clinician will receive an alert prompting them to discuss colorectal cancer screening with their patient upon visit. Patient will also receive a text message 3 days after visit reminding them to complete colorectal cancer screening.
  Arms: Arm 2B: Colonoscopy Only and Visit-Based Nudge/Text; Arm 3B: Sequential Choice and Visit-Based Nudge/Text
Behavioral: No Nudge/Text — Patient's clinician will not receive an alert prompting them to discuss colorectal cancer screening with their patient upon visit. Patient will not receive a text message 3 days after visit reminding them to complete colorectal cancer screening.
  Arms: Arm 1A: Usual Care; Arm 2A: Colonoscopy Only and No Nudge/Text; Arm 3A: Sequential Choice and No Nudge/Text

SUMMARY:
This is a 3-year pragmatic, randomized clinical trial among average-risk patients at diverse primary care practices who are overdue for colorectal (CRC) screening. This project aims to evaluate the effect of a centralized program that includes direct outreach to patients and visit-based, clinician directed nudges facilitated by the electronic health record (EHR) with follow-up text messaging on the uptake of CRC screening. The primary outcome is CRC screening completion at 3 years. Patient and clinician factors impacting the experience and effectiveness of the intervention will be explored through surveys and qualitative interviews.

DETAILED DESCRIPTION:
Despite effective strategies for prevention, early detection, and treatment, colorectal cancer (CRC) remains the second leading cause of cancer death in the United States (US). While there have been considerable policy and system-level efforts to increase CRC screening rates, uptake remains well below national goals of 80% participation. Members of racial and ethnic minorities are even further behind. Approaches to increase population-based screening can consider [1] how screening is encouraged by targeting the clinicians who typically order or recommend the procedure or the patient who completes it; and [2] the kind of screening offered (e.g., colonoscopy or fecal immunochemical testing [FIT]). This project simultaneously tests interventions along both of these dimensions.

ELIGIBILITY:
Inclusion Criteria:

* Patients ages 50-72
* Followed by Primary Care with a participating Penn Medicine PCP listed and at least one visit in the last 2 years
* Not up to date on colorectal cancer screening per Health Maintenance (no colonoscopy in the last 10 years, stool testing in the last year, flexible sigmoidoscopy in the last 5 years, MT-sDNA in the last 3 years).

Exclusion Criteria:

* Personal or significant family history of CRC, colonic polyps, hereditary nonpolyposis colorectal cancer syndrome, familial adenomatous polyposis syndrome, other gastrointestinal cancer, gastrointestinal bleeding, iron-deficiency anemia, or inflammatory bowel disease
* History of total colectomy, dementia or metastatic cancer
* Currently on hospice or receiving palliative care
* Uninsured or self-pay patients
* Currently scheduled for a colonoscopy or sigmoidoscopy
* Active order for multitarget stool DNA testing (MT-sDNA)
* History of paraplegia or quadriplegia
* Elevated chance of mortality within 3 years according to mortality risk algorithm
* Active order for Fecal Immunochemical Test (FIT) in the last 60 days
* Positive stool test (FIT or MT-sDNA) result in the last 5 years

Ages: 50 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20000 (Estimated)
Dates: Start 2023-06-07 (Actual); Primary Completion 2026-12-21 (Estimated); Study Completion 2026-12-21 (Estimated)

PRIMARY OUTCOMES:
CRC screening completion at 3 years | 3 years
  CRC screening completion at 3 years, which could be satisfied by any one of the following: colonoscopy completion at any time, negative FIT completed 2 times, or positive FIT followed by diagnostic colonoscopy within 1 year.

SECONDARY OUTCOMES:
CRC screening rate | 3 years
  CRC screening completion at 3 years by any modality
Choice of test | 3 years
  The proportion of patients who complete CRC screening by screening type

CONTACTS AND LOCATIONS:
Overall Officials: Shivan Mehta, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Penn Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mehta SJ, Shaw PA, Reitz C, Brophy C, Okorie E, Williams K, Segura A, Tao J, Snider CK, Wollack C, Friday S, Rendle KA, Klaiman T, Glanz K, Rhodes C, Asch DA. Sequential choice vs colonoscopy outreach for colorectal cancer screening: Design and rationale of a pragmatic randomized clinical trial. Contemp Clin Trials. 2025 Dec 16;161:108188. doi: 10.1016/j.cct.2025.108188. Online ahead of print. PMID 41412475